CLINICAL TRIAL: NCT01627834
Title: Open Label, Balanced, Randomized, Two-treatment, Two-sequence, Two-period, Single-dose, Crossover Oral Bioequivalence Study of Ropinirole Hydrochloride Extended Release Tablets 2 mg of Dr. Reddy's Laboratories Limited, India With REQUIP@ XL (Ropinirole) 2 mg ER Tablets of Glaxosmithkline, USA, in Normal, Healthy, Adult, Human Subjects Under Fasting Condition.
Brief Title: Bioequivalence Study of Ropinirole Hydrochloride ER Tablets 2 mg Under Fasting Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 034-09
Record Dates: First submitted 2012-06-22; First posted 2012-06-26 (Estimated); Last update posted 2012-09-28 (Estimated); Status verified 2010-01

CONDITIONS: Healthy
Keywords: Bioequivalence; Ropinirole Hydrochloride; crossover
MeSH Terms: interventions — ropinirole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ropinirole (Experimental): Ropinirole Hydrochloride ER tablets 2 mg of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Ropinirole
- Requip (Active Comparator): Requip XL Tablets 2 mg of Glaxosmithkline, USA
  Interventions: Drug: Ropinirole

INTERVENTIONS:
Drug: Ropinirole
  Other Names: Requip

SUMMARY:
This is an open label, randomised, balanced, two-treatment, two-period, two-sequence, crossover, oral bioequivalence study.

DETAILED DESCRIPTION:
The objective of this study was to determine the single-dose oral bioequivalence of Ropinirole Hydrochloride Extended Release Tablets 2 mg of Dr. Reddy's Laboratories Limited, India with REQUIP® XL (Ropinirole) 2 mg ER Tablets of Glaxosmithkline, USA, in normal, healthy, adult, human subjects under fasting condition.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy human subjects aged between 18 and 45 years (including both).
2. Subjects with a BMI between 18.5 - 24.9 Kg/m2 (including both) but body weight not less than 45 Kgs.
3. Subjects with normal health as determined by personal medical history, clinical examination, and laboratory examinations including serological tests.
4. Subjects having normal 12-lead electrocardiogram (ECG).
5. Subjects having normal chest X-Ray (PIA view).
6. Subjects able to communicate effectively.
7. Subjects willing to give written informed consent and adhere to all the requirements of this protocol.
8. Female subjects who are postmenopausal or surgically sterile.
9. Female subjects practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies, diaphragm,intrauterine device (IUD) or abstinence.

Exclusion Criteria:

1. Subjects having contraindications or hypersensitivity to ropinirole or domperidone or related group of drugs.
2. History or presence of any medical condition or disease according to the opinion of the physician.
3. History or presence of significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological, neurological or psychiatric disease or disorder.
4. History or presence of significant alcoholism or drug abuse in the past one year.
5. History or presence of significant smoking (more than 10 cigarettes or bidis/day or consumption of tobacco products).
6. Difficulty with donating blood.
7. Difficulty in swallowing solids like tablets or capsules.
8. Systolic blood pressure less than 110mm Hg or more than 140 mm Hg.
9. Diastolic blood pressure less than 70 mm Hg or more than 90 mm Hg.
10. Pulse rate less than 50 beats/minute or more than 100 beats/minute.
11. Use of any prescribed medication during last two weeks or OTC medicinal products during the last one week preceding the first dosing.
12. Major illness during 3 months before screening.
13. Participation in a drug research study within past 3 months.
14. Donation of blood in the past 3 months before screening.
15. Female subjects demonstrating a positive pregnancy screen.
16. Female subjects who are currently breast-feeding.
17. Female subjects with child bearing potential using prohibited contraceptive method (Oral, Injectable or Implantable hormonal agents).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2009-10; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Area under curve(AUC) | Pre-dose (before dosing, in the morning of the day of dosing) and at 1.00, 2.00, 3.00,4.00, 5.00, 6.00, 7.00, 8.00, 9.00, 10.00, 11.00, 12.00, 13.00, 14.00, 15.00, 16.00, 17.00, 18.00,20.00, 24.00, 30.00, 36.00, 48.00 and 60.00 hours after dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Naba Kr Talukdar, MD, Principal Investigator — GVK Biosciences Pvt. Ltd.
Locations (1):
- GVK Biosciences Pvt. Ltd, Ameerpet, Hyderabad, India